CLINICAL TRIAL: NCT03898388
Title: A Prospective Analysis Correlating the Osteoarthritic Knee Microenvironment to Clinical Outcome After Treatment With Regenexx® SD Treatment: A Multi-Site Study
Brief Title: Correlating the OA Knee Microenvironment to Outcomes After Regenexx-SD Treatment: A Multi-Site Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor discontinued study-impacted by COVID
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGX2018-LAB01
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee Synovial Fluid collection before Regenexx-SD (Experimental): Measure components of knee synovial fluid 2-4 days before the Regenexx-SD treatment.
  Interventions: Procedure: Bone Marrow Concentrate treatment

INTERVENTIONS:
Procedure: Bone Marrow Concentrate treatment — Correlate patient outcomes 6 months after receiving the Regenexx SD treatment with measurements of synovial fluid collected before treatment
  Other Names: Regenexx®SD Treatment

SUMMARY:
Multi-center study to include up to 600 subjects with knee osteoarthritis in unilateral or bilateral knees treated with Regenexx® SD in the osteoarthritic knee/s. Synovial fluid drawn from patients' knee/s prior to receiving Regenexx-SD treatment will be correlated with their clinical outcomes after treatment.

DETAILED DESCRIPTION:
Initial study procedures include baseline evaluation of medical history, knee history, knee examination, medication use, MRI, and subject-reported outcomes.

Each osteoarthritic subject will undergo withdrawal of knee joint synovial fluid for each knee being treated (0.3-0.5 ml) which will be analyzed by the research laboratory via multiplexed enzyme linked immunosorbent assay (ELISA) and dimethylmethylene blue assay (DMMB) at pre-injection (2-8 days before Regenexx-SD treatment). Documentation of osteoarthritic joint characteristics and injection procedure details will be recorded throughout the study.

The unaffected knee joint will undergo no treatment, but bilateral knees may be treated.

The objective of this study is to correlate the pre- Regenexx-SD treatment levels of pro-inflammatory cytokines, anti-inflammatory cytokines, matrix metalloproteinases, and catabolic articular cartilage breakdown products in the osteoarthritic knee synovial fluid microenvironment with 6 month post-treatment clinical outcomes. This data will be used to establish a predictive a priori testing "model" to determine if a patient is a good candidate for the Regenexx-SD treatment based on their initial osteoarthritic knee synovial fluid microenvironment phenotype. It may also be used to determine if the micro-environment can be altered to improve outcome before receiving Regenexx-SD.

Incidence of post-operative complications, adverse events, re-injections, and surgical intervention and change in pain score will be considered while determining these direct and indirect associations upon completion of the Regenexx-SD treatment.

Components of the synovial fluid will be correlated to post-treatment clinical outcomes, which include several self-reported questionnaires as well as assessment of post-injection complications, adverse events, re-injections and surgical interventions. Patient reported questionnaires include IKDC Subjective Knee Evaluation, Lower Extremity Function Scale, Pain Scales and a Modified Single Assessment Numeric Evaluation (SANE).

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary signature of the IRB approved Informed Consent 2) Unilateral or bilateral osteoarthritic male or female ages 35-85 3) Pain, swelling, and/or functional disability in the affected knee consistent with osteoarthritis in the knee joint 4) Physical examination consistent with osteoarthritis in one knee joint 5) Kellgren-Lawrence grade 2 or greater knee osteoarthritis and/or diagnostic MRI imaging of the affected knee showing osteoarthritis (i.e. chondral loss, fissuring, defect, bone marrow lesion, meniscus tear, synovial thickening, etc.) 6) Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

* 7) Knee injections of any type within 3 months prior to the study. 8) Knee surgery within 6 months prior to the study.

  9) Patient undergoing lavage with treatment

  10) Inflammatory or auto-immune based joint diseases or other lower extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout) 11) Quinolone or statin-induced myopathy/tendinopathy 12) Severe neurogenic inflammation of the cutaneous nerves about the knee or thigh 13) Contraindications for MRI 14) Condition represents a worker's compensation case 15) Currently involved in a health-related litigation procedure 16) Is pregnant 17) Bleeding disorders 18) Currently taking anticoagulant or immunosuppressive medication 19) Allergy or intolerance to study medication 20) Use of chronic opioid 21) Documented history of drug abuse within six months of treatment 22) Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Correlation between components in knee synovial fluid to patient-reported outcomes post-procedure. | 6 months after Regenexx-SD treatment
  1) Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to IKDC delta scores at 6 months.

SECONDARY OUTCOMES:
Correlation between components of synovial fluid to 12 month IKDC outcomes | 12 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to IKDC delta scores at 12 months.
Correlation between components of synovial fluid and 6 month pain score | 6 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to pain scale deltas at 6 months.
Correlation between components of synovial fluid and 6 month Lower Extremity Function Scale (LEFS). | 6 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to LEFS deltas at 6 months.
Correlation between components of synovial fluid and 6 month modified Single Assessment Numeric Evaluation (SANE) | 6 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to SANE scores at 6 months.
Correlation between components of synovial fluid and 12 month pain scores | 12 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to pain scale deltas at 12 months.
Correlation between components of synovial fluid and 12 month LEFS | 12 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to LEFS deltas at 12 months.
Correlation between components of synovial fluid and modified SANE | 12 months
  Correlations between cytokine levels, matrix metalloproteinase levels, and catabolic cartilage breakdown products from pre-treatment synovial fluid to modified SANE scores at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Regenexx, LLC
Locations (3):
- United States (3):
  - Interventional Orthopedics of Atlanta, Atlanta, Georgia
  - Regenexx Des Moines, Des Moines, Iowa
  - Regenexx Las Vegas, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centeno CJ, Al-Sayegh H, Bashir J, Goodyear S, Freeman MD. A dose response analysis of a specific bone marrow concentrate treatment protocol for knee osteoarthritis. BMC Musculoskelet Disord. 2015 Sep 18;16:258. doi: 10.1186/s12891-015-0714-z. PMID 26385099
- [Background] Centeno C, Sheinkop M, Dodson E, Stemper I, Williams C, Hyzy M, Ichim T, Freeman M. A specific protocol of autologous bone marrow concentrate and platelet products versus exercise therapy for symptomatic knee osteoarthritis: a randomized controlled trial with 2 year follow-up. J Transl Med. 2018 Dec 13;16(1):355. doi: 10.1186/s12967-018-1736-8. PMID 30545387
- [Background] Themistocleous GS, Chloros GD, Kyrantzoulis IM, Georgokostas IA, Themistocleous MS, Papagelopoulos PJ, Savvidou OD. Effectiveness of a single intra-articular bone marrow aspirate concentrate (BMAC) injection in patients with grade 3 and 4 knee osteoarthritis. Heliyon. 2018 Oct 18;4(10):e00871. doi: 10.1016/j.heliyon.2018.e00871. eCollection 2018 Oct. PMID 30364761
- [Background] Centeno CJ, Al-Sayegh H, Freeman MD, Smith J, Murrell WD, Bubnov R. A multi-center analysis of adverse events among two thousand, three hundred and seventy two adult patients undergoing adult autologous stem cell therapy for orthopaedic conditions. Int Orthop. 2016 Aug;40(8):1755-1765. doi: 10.1007/s00264-016-3162-y. Epub 2016 Mar 30. PMID 27026621